CLINICAL TRIAL: NCT06873893
Title: Efficacy of Ultrasound Guided Pectoral Nerve Block Versus Ultrasound Guided Mid-point Transverse Process Block for Postoperative Analgesia in Patients Undergoing Modified Radical Mastectomy
Brief Title: Comparing Between Ultrasound Guided Pectoral Nerve Block Versus Ultrasound Guided Mid-point Transverse Process Block for Postoperative Analgesia in Patients Undergoing Modified Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmin tarek ali ahmed elshahawy, Assistant lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD11/2024
Record Dates: First submitted 2025-02-16; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pectoral nerve block group (Active Comparator): This group will receive a volume of 10ml of bupivacaine 0.5% will be injected between the pectoralis major and pectoralis minor muscle then another 10ml bupivacaine will be injected between pectoralis minor and serratus anterior muscle
  Interventions: Procedure: Pectoral Nerve Block
- Mid-point transverse process block group (Active Comparator): This group will receive a volume of 20ml of bupivacaine 0.5% at midpoint of the line between the posterior border of the transverse process of T4 and the pleura ( injection will be deep to the posterior aspect of the vertebral transverse process but superficial to the superior costotransverse ligament )
  Interventions: Procedure: Midpoint transverse process block

INTERVENTIONS:
Procedure: Midpoint transverse process block — This group will receive a volume of 20ml of bupivacaine 0.5% at midpoint of the line between the posterior border of the transverse process of T4 and the pleura ( injection will be deep to the posterior aspect of the vertebral transverse process but superficial to the superior costotransverse ligament )
  Arms: Mid-point transverse process block group
Procedure: Pectoral Nerve Block — This group will receive a volume of 10ml of bupivacaine 0.5% will be injected between the pectoralis major and pectoralis minor muscle then another 10ml bupivacaine will be injected between pectoralis minor and serratus anterior muscle
  Arms: pectoral nerve block group

SUMMARY:
The aim of the study is to compare the effectiveness of ultrasound guided pectoral nerve block versus mid-point transverse process block for postoperative analgesia in patients undergoing modified radical mastectomy

DETAILED DESCRIPTION:
preoperative assessment will be done for every patient including history, clinical examination &laboratory investigation ( coagulation profile ) according to age , physical state . all patients will be instructed about numeric rating scale of pain (NRS) , intravenous access will be placed under complete aseptic condition . on arriving to operating room , standard ASA monitoring ( ECG , non invasive arterial blood pressure and pulse oximetry ) will be assembled. baseline readings of all vital data will be recorded before induction , induction of anesthesia will be done by propofol 2mg/kg , atracurium 0.5mg/kg and fentanyl 1mcg/kg . endotracheal intubation will be placed then patients will be mechanically ventilated with setting keeping end tidal CO2 between 35-45 mmHg . anesthesia will be maintained with volatile anesthetic (isoflurane) and atracurium 0.1mg/kg every 20 minutes, maintenance fluid will be given according to patient's weight , fasting hours , and duration of surgery . incremental doses of fentanyl ( 1mcg/kg ) will be given every 2 hours according to duration of surgery . all patients will receive 1gm parecetamol with skin closure .

both blocks will be done by an experienced anesthesiologist in sonar guided peripheral nerve blockade under complete aseptic conditions, after induction of general anesthesia .

patients will be randomly divided into two groups P-Group : pectoral nerve block patient will be positioned in supine position and patient's arm next to the body , the linear probe (10-12 MHz) will be positioned in the parasagittal plane below the lateral half of the clavicle . the pectoral branch of the thoraco-acromial artery will be identified between pectoralis major and minor using color doppler. in-plane needle approach will be used , and the needle will be advanced from medial to lateral direction enter the plane between pectoralis major and pectoralis minor , a volume of 10ml of bupivacaine 0.5% will be injected between the two muscles (the interpectoral plane ) with careful intermitted aspiration to avoid intravascular injection . Then the needle will be advanced into the plane between te pectoralis minor and serratus muscles , and 10ml of bupivacaine will be injected watching for the spread between two muscles under ultrasound guidance with careful intermitted aspiration to avoid intravascular injection M-Group : mid-point transverse process block in the lateral position , the T4 spine will be counted by ultrasound and high frequency linear probe (10-12MHz) will be placed longitudinally , approximately 2.5 cm lateral to the midline the needle will be advanced in plane from cranial to caudal direction , the desired end point for the needle tip will be the midpoint of the line between the posterior border of transverse process of T4 and the pleura (injection will be deep to the posterior aspect of the vertebral transverse process but superficial to the superior costotransverse ligment) the needle tip does not enter the paravertebral space , a volume of titrated bolus of 20ml of bupivacaine 0.5% will be injected after aspiration to avoid intravascular injection, pleural displacement and bowing of erector spinae will be observed at the side of injection

ELIGIBILITY:
Inclusion Criteria:

* all female patients undergoing modified radical mastectomy
* age between 35 to 65

Exclusion Criteria:

* patient refusal of procedure or participation in the study
* duration of operation more than 180 minutes
* known ASA IV or more
* local skin infection at site of the block
* contraindication of local anesthetic infiltration ( history or evidence of coagulopathy , use of anticoagulant or antiplatelet therapy , known allergy of local anethestic (bupivacaine )

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the time to first rescue analgesia for every patient | Up to 18 hours after surgery , time between end of operation and when patients ask for rescue analgesia with NRS 4 or more
  when the patients with numeric rating scale 4 or more will receive 5mg morphine IV as rescue analgesia (the higher numeric rate score means a worse outcome)

SECONDARY OUTCOMES:
-Number of patients requested rescue analgesia | 18 hour postoperative
The total number of doses of rescue analgesia | 18 hours postoperatively
  -the total number of doses of rescue analgesia that will be administered in the 18 hours postoperatively if the NRS pain score at rest 4 or more
Incidence of complications | 18 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo , Abbassya, Egypt

IPD SHARING:
Plan to Share IPD: No